CLINICAL TRIAL: NCT00308646
Title: Instrument Development of Screening Prediabetes Patients
Status: Terminated | Type: Observational
Sponsor: China Medical University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: NSC93-2314-B-039-025
Record Dates: First submitted 2006-03-29; First posted 2006-03-30 (Estimated); Last update posted 2006-03-30 (Estimated); Status verified 2006-03

CONDITIONS: Prediabetic State
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
It will be more effective if we can work on the primary prevention for the high risk groups of diabetes and prediabetes such as the early detection.

DETAILED DESCRIPTION:
During the past years, many efforts were put on the diagnosis and treatment of DM and its complications. It will be more effective if we can work on the primary prevention for the high risk groups of diabetes and prediabetes such as the early detection. As a first public health step, it is worthwhile to identify prediabetes people in community by screening program. Three thousand persons will be randomly selected from residents of Taichung city. All the participants will fulfill a structured questionnaire and 'Diabetes risk factor screening tool' which American Diabetes Association suggested in 2003. This project will estimate the prevalence of prediabetes in conventional hospital-base population as well as the validity of a screening questionnaire for prediabetes.

ELIGIBILITY:
Inclusion Criteria:

Residents aged 40 and over of Taichung city, Taiwan in October, 2004.

Exclusion Criteria:

-

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000
Dates: Start 2004-10; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Lin C Chieh, Professor, Principal Investigator — School of Medicine, China Medical University